CLINICAL TRIAL: NCT04599257
Title: Simultaneous Application of High-Intensity Focused Electromagnetic Procedure and Radiofrequency for Changes in Subcutaneous Fat Tissue and Muscle Toning of Thighs
Brief Title: Fat Reduction and Muscle Toning of Thighs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-703_300
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Fat Burn
Keywords: muscle strengthening; muscle tone; fat reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hip and thigh circumference changes (Experimental): The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete four (4) treatment visits and two to three follow-up visits. All of the study subjects will receive the treatment with the subject device.
  At the baseline visit, MRI imaging will be performed; the subject's weight and hip and thigh circumference will be recorded. Photos of the treated area will be taken.
  The treatment administration phase will consist of four (4) treatments, delivered once a week. The applicator of the device will be applied over the treatment area. The device will induce visible muscle contractions along with heating of the subcutaneous fat.
  At the last therapy visit, the subject's weight and hip and thigh circumference will be recorded, and photos of the treated area will be taken. In addition, subjects will receive Subject Satisfaction Questionnaire to fill in.
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — The device applicator combines high-intensity focused electromagnetic procedure and radiofrequency energy to induce visible muscle contractions along with heating of the subcutaneous fat.

SUMMARY:
This study will evaluate the clinical efficacy and safety of a simultaneous application of high-intensity focused electromagnetic procedure and radiofrequency energy for changes in subcutaneous fat tissue and muscle toning of thighs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Voluntarily signed an informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain her regular (pre-procedure) diet and exercise regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Injured or otherwise impaired muscles
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, nursing, and menstruation
* Intrauterine device (IUD)
* Swollen or neoplastic tissues, space-occupying lesions or skin eruptions in the treatment area
* Basedow's disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of structural changes of subcutaneous tissues between pre-treatment and post-treatment based on MRI imaging | 7 months
  The primary objective of the study is to determine the effectiveness of a simultaneous application of high-intensity focused electromagnetic procedure and radiofrequency energy for change in the adipose layer thickness between pre-treatment and post-treatment based on MRI imaging. The changes will be considered statistically significant where p-value <0.05.

SECONDARY OUTCOMES:
Assess subjects' satisfaction with the treatment using Subject Satisfaction Questionnaire | 7 months
  The 5-point Likert scale Satisfaction questionnaire will be used to evaluate the participant's satisfaction with the therapy outcome. Subject satisfaction will be assessed after the last therapy visit and during the follow-up visits with 4-therapy related questions with answer "Strongly agree" will be the best possible answer and "Strongly disagree" the worst.
Assess safety profile by recording of adverse events | 7 months
  All AEs including local and systemic reactions not meeting the criteria for "serious adverse events" will be captured on the appropriate CRF. Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product (assessed only by those with the training and authority to make a diagnosis, which would include MD, DDS, DMD, PA, Nurse Practitioner or DO), and time of resolution/stabilization of the event. All AEs occurring during the study must be documented appropriately regardless of relationship to study device. All AEs will be followed to adequate resolution.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Brian M. Kinney M.D., Inc, Beverly Hills, California
  - Art of Skin MD, Solana Beach, California
  - Yael Halaas, M.D., F.A.C.S., New York, New York
  - Center For SmartLipo & Plastic Surgery, Langhorne, Pennsylvania

IPD SHARING:
Plan to Share IPD: No